CLINICAL TRIAL: NCT01090973
Title: Phase II Trial of Oral LBH 589, a Novel Histone Deacetylase (HDAC) Inhibitor, in Relapsed or Refractory Chronic Lymphocytic Leukemia and Mantle Cell Lymphoma
Brief Title: Oral LBH589 in Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) and Mantle Cell Lymphoma (MCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company request.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15971; IRB # Pro00000102 (Other: USF Institutional Review Board); CLBH589B25T (Other: Novartis)
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: relapsed; refractory; CLL; chronic lymphocytic leukemia; MCL; mantle cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — Panobinostat; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral drug treatment (Experimental): LBH589 will be given orally (by mouth), 40 mg once-a-day, 3 times weekly every week on days 1, 3 & 5, then 8, 10 &12, then 15, 17 & 19, then 22, 24 & 26.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — The LBH589 capsule(s) should be swallowed by mouth with a glass of water (8 ounces noncarbonated) in the morning. The daily dose of LBH589 should be taken at approximately the same time each day. Patients should avoid eating grapefruit, Seville (sour) orange or drinking grapefruit juice or Seville orange juice during the study.
  After 2 cycles of treatment, if patients do not demonstrate a partial response or complete response (all of the tumor is gone) to the therapy they will be removed from the study. If patients do obtain a partial (the tumor(s) have decreased in size or number but there are still tumors present) or complete response then treatment will continue until their disease progresses.
  Other Names: panobinostat; HDAC Inhibitor

SUMMARY:
The purpose of the study is to find out the effects and the safety of an investigational study drug called LBH589 when given to people with relapsed or refractory chronic lymphocytic leukemia (CLL) or mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
Response Assessment for Mantle Cell Lymphoma

Based on the International Workshop to Standardize Response Criteria to non-hodgkin's lymphoma (NHL) (Cheson, JCO 1999) a complete hematologic remission will be defined as the following:

* Disappearance of all evidence of disease.
* Any positron emission tomography (PET)+ mass prior to therapy must be PET negative after treatment.
* No palpable spleen or liver
* If bone marrow involvement prior to therapy, must document clear bone marrow.

Partial response will be defined as:

* No new areas of disease on clinical exam and regression of previous areas of disease
* Greater than or equal to 50% decrease in the size of prior disease areas per measurement on computed tomography (CT) scan
* No new PET+ areas on PET scan
* No increase in size of liver or spleen

Response Assessment for CLL

Using the National Cancer Institute (NCI) criteria, a complete hematologic remission will be defined as having the following present for 2 or more months:

* Absence of symptoms attributable to CLL
* Normal findings on physical examination
* Absolute lymphocyte count <4000/microL
* Absolute neutrophil count (ANC) >1500/microL
* Platelet count >100,000/microL
* Hemoglobin concentration >11 g/dL (untransfused)
* Bone marrow lymphocytosis <30 percent
* No nodules (lymphoid aggregates) on bone marrow biopsy

A partial response per the NCI criteria will be defined as having the following for 2 or more months:

* A reduction in previously enlarged nodes, spleen, and liver by at · least 50 percent and
* Absolute neutrophil count ≥1500/microL or
* Platelet count ≥100,000/microL or
* Hemoglobin concentration ≥11 g/dL or
* 50 percent improvement over pretherapy reductions in hemoglobin concentration and/or platelet count

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Patients must meet the following laboratory criteria (unless dysfunction is due to organ infiltration by lymphoma):

  * ANC ≥ 1.5 x 10^9/L
  * Hemoglobin ≥ 9 g/dl
  * Platelets ≥ 75 x 10^9/L
  * Calculated CrCl ≥50 mL/min (MDRD Formula)
  * Total serum calcium ≥ LLN
  * Total serum magnesium ≥ LLN
  * Aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN
  * Serum bilirubin ≤1.5 x ULN
  * Serum potassium ≥ LLN
  * Thyroid stimulating hormone (TSH) ≥ lower limit of normal (LLN) and free T4 within normal limits. Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Baseline multiple uptake gate acquisition scan (MUGA) or echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional normal.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Documented MCL by biopsy or CLL by biopsy or flow cytometry.
* Relapsed or refractory disease despite 1 or more lines of therapy.

Exclusion Criteria:

* Prior histone deacetylase (HDAC), DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Peripheral neuropathy ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 3
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * Patients with congenital long QT syndrome
  * History or presence of sustained ventricular tachyarrhythmia. (Patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
  * History of ventricular fibrillation or torsade de pointes
  * Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
  * Screening 12 lead electrocardiogram (ECG) with a QTc > 450 msec
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
  * Other clinically significant heart disease (e.g., congestive heart failure (CHF) New York Heart Association (NYHA) class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LBH589
* Patients with diarrhea > CTCAE grade 1
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (which ever is longer) and who have not recovered from side effects of those therapies.
* Have received either immunotherapy within < 8 weeks; chemotherapy within < 4 weeks; or radiation therapy to > 30% of marrow-bearing bone within < 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
* Have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). WOCBP must have a negative serum pregnancy test within 24 hours of receiving the first dose of study medication.
* Male patients whose sexual partners are WOCBP not using effective birth control
* Prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
* Have not received prior therapy for aggressive MCL or CLL.
* No documentation of disease refractoriness (i.e. progression of disease despite current therapy or recurrence within 3 months of last treatment) or relapse despite prior therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Bello, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Drug Treatment: LBH589 was to be given orally (by mouth), 40 mg once-a-day, 3 times weekly every week on days 1, 3 & 5, then 8, 10 &12, then 15, 17 & 19, then 22, 24 & 26.
Period: Overall Study
Arm/Group | Oral Drug Treatment
Started | 1
Completed | 0
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Desired Response
Description: Investigators intended to assess the rate of overall and complete response by World Health Organization (WHO) classification in patients with relapsed or refractory aggressive mantle cell lymphoma (MCL) and chronic lymphocytic leukemia (CLL).
  WHO Performance Scale Measures levels of patient capability: 0 Normal activity; 1 Symptoms, but nearly fully ambulatory; 2 Some bed time, but needs to be in bed <50% of normal daytime; 3 Needs to be in bed >50% of normal daytime; 4 Unable to get out of bed.
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: The study was abandoned after only one patient due to low accrual and the sponsor losing interest in the single-agent.
  The one patient had disease progression requiring more aggressive treatment and did not complete the study.
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Complete Response (CR) and Partial Response (PR)
Description: Investigators intended to determine the complete and partial responses. Chronic Lymphocytic Leukemia (CLL): Using the NCI criteria - - See definitions in the Detailed Description section for a Complete hematologic Remission, and Partial Response.
  Mantle Cell Lymphoma (MCL): Based on the International Workshop to Standardize Response Criteria to NHL (Cheson, JCO 1999) - See definitions in the Detailed Description section for a Complete hematologic Remission, and Partial Response.
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: as for outcome 1
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Response Duration
Description: Investigators intended to determine the duration of responses.
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: as for outcome 1
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS) Estimate
Description: Investigators intended to estimate the progression free survival time
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: as for outcome 1
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Prolonged Corrected QT (QTc) Interval
Description: Investigators intended to monitor the QTc interval in patients receiving oral LBH589
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Improved Blood and Lymphatic Evaluation Results
Description: Investigators intended to evaluate histone acetylation, cytotoxic mixed lymphocyte reaction (MLR) activity, cytokine profiles, and immunologic synapse alterations through peripheral blood correlative studies
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: as for outcome 1
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Investigators intended to evaluate the safety and tolerability profile of LBH589. Assessments would consist of monitoring and recording all adverse events and serious adverse events, the regular monitoring of hematology, blood chemistry and urine values, vital signs, ECOG performance status, and the regular physical examinations and ECG assessments.
  Adverse events will be assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 3.0. CTCAE v3.0 can be accessed on the National Institute of Health (NIH)/NCI website at http://ctep.cancer.gov/forms/CTCAEv3.pdf.
Time Frame: 8 weeks (2 cycles) unless treatment continues due to partial or complete response
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Oral Drug Treatment
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 46 days
Arm/Group | Oral Drug Treatment
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Drug Treatment (N=1)
Death not associated with CTCAE term - Disease progression NOS (Blood and lymphatic system disorders) | 1 (1) — Grade 5. Unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Drug Treatment (N=1)
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1 (1) — Grade 3. Unrelated to study drug.

LIMITATIONS AND CAVEATS:
The study was abandoned after only one patient due to low accrual and the sponsor losing interest in the single-agent.

The one patient had disease progression requiring more aggressive treatment and did not complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes